CLINICAL TRIAL: NCT02087267
Title: Lumbar Fusion With The Icotec CF/PEEK Pedicle System In Combination With The Icotec CF/PEEK TLIF Cage ETurn™
Status: Completed | Type: Observational
Sponsor: Sitona AG (Other)
Responsible Party: Sponsor
Other Study IDs: SITONA_01/2014
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Degeneration of Lumbar Intervertebral Disc; Degenerative Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1- or 2-level spinal fusion: Patients suffering from symptomatic degenerative disc disease or degenerative spondylolisthesis grade 1 or 2 with chronic low back pain, pain in the leg or buttock, muscle weakness, sensation abnormalities and/or neurogenic claudication requiring 1- or 2-level lumbar or lumbar-sacral spinal fusion.
  Interventions: Procedure: 1- or 2-level spinal fusion

INTERVENTIONS:
Procedure: 1- or 2-level spinal fusion — 1- or 2-level lumbar or lumbar-sacral spinal fusion with the icotec CF/PEEK Pedicle System in combination with the icotec CF/PEEK TLIF Cage ETurn™

SUMMARY:
The objective of the PMCF is to collect outcome information on patients suffering from symptomatic degenerative disc disease or degenerative spondylolisthesis requiring 1- or 2-level lumbar or lumbar-sacral spinal fusion with posterior instrumentation and therefore receiving the icotec CF/PEEK Pedicle System in combination with the icotec CF/PEEK TLIF Cage ETurn™.

DETAILED DESCRIPTION:
Background: At present, metal pedicle screw systems made from titanium or stainless steel are commonly used for posterior stabilization. One disadvantage of theses metal devices is that they cause shadows and artifacts on CTs and MRIs which may hamper the postoperative exploration of the onset of spinal diseases and in particular the evaluation of the neuroforamina, the spinal canal and bone-implant interfaces. Therefore new concepts of pedicle screw devices use non-radiopaque materials such as carbon fiber-reinforced polyetheretherketone (CF/PEEK) without compromising mechanical properties compared to standard titanium implants and possibly reducing the risk for adjacent segment diseases.

Description of the study devices:

The icotec Pedicle System is intended to provide immobilization and stabilization of spinal segments in skeletally mature patients as an adjunct to fusion in the treatment of acute and chronic instabilities or deformities of the thoracic, lumbar and sacral spine. The carbon fiber-reinforced polyetheretherketone (CF/PEEK) that is used to produce the icotec pedicle system rod and screw shaft is a thermoplastic composite biomaterial exhibiting properties suitable for load-bearing orthopedic implants. The CF/PEEK material does not cause artifacts or shadows on adjacent tissues with all imaging modalities such as x-ray, CT, and MRI. Radiopaque markers or fibres made from titanium or tantalum are embedded. The pedicle system rod and screws allow this advantage to be realized without compromising mechanical properties compared to standard titanium implants.

Description of the study device - icotec CF/PEEK TLIF Cage ETurn: The icotec ETurn™ TLIF cage consists of a windowed body with a central slot, a distraction/ insertion wedge and surface treads on its cranial and caudal surfaces that serve to guide and anchor the implant (see figure 4). The concentrically arranged treads enable the implant to turn on its own from its position of insertion into the disc space to its transverse end position. The tread surfaces help to create a significantly larger pressure-bearing contact surface between the implant and the bone than the conventional pointed anchoring elements.

Risk Analysis and risk Management: Most of the risks of implant related, surgical and postoperative complications associated with the implantation of the icotec CF/PEEK Pedicle System in combination with the icotec ETurn™ TLIF cage, are comparable to the risks associated with other TLIF surgeries with cages and pedicle screw systems intended for lumbar spine stabilization.

risks and possible adverse outcomes have been identified for the icotec CF/PEEK Pedicle System as well as for the CF/PEEK TLIF Cage ETurn.

Legal Aspects: For this post-market investigation only CE-marked medical devices will be used within their intended purpose and no additional invasive or other stressful examinations are to be carried out.

All subjects will voluntarily sign the Informed Consent document. Ethics approval for the study will be obtained prior to starting the study

Data Monitoring: Independent on-site Monitoring will be performed at all investigational sites.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic degenerative disc disease or degenerative spondylolisthesis grade 1 or 2 with chronic low back pain, pain in the leg or buttock, muscle weakness, sensation abnormalities and/or neurogenic claudication
* Unsuccessful adequate conservative treatment
* 1- or 2- contiguous level lumbar spinal fusion between L2 and S1 with posterior instrumentation in combination with Transforaminal Lumbar Interbody Fusion (TLIF)
* Age between 18 - 80 years at the time of surgery
* Skeletally mature patient
* Patient understands the conditions of the study and is willing and able to comply with the postoperative scheduled clinical and imaging evaluations and the prescribed rehabilitation
* Patient signed Informed Consent

Exclusion Criteria:

* No adequate non-operative care prior to being treated with a lumbar fusion device
* 3-level fusion or more
* Fusion not between L2 and S1
* Previous lumbar spinal surgery, other than discectomy at the level(s) to be operated on
* Spondylolisthesis acc. to Meyerding grade 3 or higher
* Transforaminal access to the disc space is obstructed
* Use of bone grafts other than autologous grafts, demineralized bone matrix without additional growth factors and synthetic bone substitute without additional growth factors. Growth factor enhanced grafts, cement or any other graft material are excluded.
* Adiposity, severe obesity (BMI > 35 kg/m2)
* Any contraindication for MRI scan including heart pacemaker, metallic foreign body (metal sliver) in the eye or brain, aneurysm clip in the brain, severe claustrophobia etc.
* Discitis, spondylodiscitis
* Acute or chronic infection, previous surgical site infection or severe defect of the osseous structures
* Open wounds
* Patient who takes immunosuppressive or long-term steroid use
* Fever
* Allergy or intolerance to any device material (e.g. Carbon/PEEK, titanium or tantalum)
* Foreign body sensitivity
* Insufficient form fit between the implant and the bone owing to deformation or destruction of the pedicles or of the vertebral body end plates
* Risk that the intervertebral device can subside into the vertebral bodies
* Bone tumors in the region of the implant anchoring
* Severe osteoporosis or similar bone density loss, incl. any metabolic bone disease
* Cases, in which the progression of degenerative disease is so advanced at the time of implantation that it may substantially decrease the expected useful life of the appliance
* Systemic or metabolic illnesses (i.e. insulin-dependent diabetes)
* Patient who is suffering from rheumatological or other inflammatory joint disease
* Paralysis of lower extremity
* Generally poor condition of the patient
* Psychosocial issues; lack of co-operation by the patient
* Drug abuse or alcoholism
* Any medical or surgical condition that could preclude the potential success of the implantation
* Any condition not described in the indications for use
* Unwillingness or inability of the patient to follow the instructions for postoperative treatment or with the follow-up evaluation schedule
* Female patient who is pregnant or plans to become pregnant during the course of the study
* Prisoner
* Patient who has not signed the Informed Consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic of selected spine centers
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Overall fusion rate | 2 years postoperatively
  Outcome Measure by CT/MRI and clinical follow-up

SECONDARY OUTCOMES:
Rate of pedicle system implant failures | 2 years postoperatively
  Outcome Measure by CT/MRI and clinical follow-up
Rate of implant related, surgery related, postoperative and general complications | 2 years postoperatively
  Outcome Measure by CT/MRI and clinical follow-up
Rate of subsequent surgical interventions | 2 years postoperatively
  Outcome Measure by CT/MRI and clinical follow-up
Change of the mean total Oswestry Low Back Pain Disability Questionnaire (ODI) | Change from the preoperative baseline to the 2 year postoperative assessment
  clinical follow-up
Change of the mean Visual Analogue Scale (VAS) on low back pain | Change from the preoperative baseline to the 2 year postoperative assessment
  clinical follow-up
Change of the mean Visual Analogue Scale (VAS) on pain in the leg and buttock (experienced in the pain-dominant leg) | Change from the preoperative baseline to the 2 year postoperative assessment
  clinical follow-up
Visual Analogue Scale (VAS) on patient's satisfaction with the surgery | 2 years postoperatively
  clinical follow-up
Change of the mean disc height at index level | Change from the preoperative baseline to the 2 year postoperative assessment
  Outcome Measure by CT/MRI and clinical follow-up
Rate of symptomatic adjacent segment disease | 2 years postoperatively
  Outcome Measure by CT/MRI and clinical follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Eif, MD, Principal Investigator — Städtisches Klinikum Görlitz gGmbH
Locations (6):
- Germany (5):
  - Universitätsklinikum SH Klinik für Neurochirurgie, Kiel, Schleswig-Holstein
  - Orthopädische Universitätsklinik Friedrichsheim gGmbH, Frankfurt am Main
  - Städtisches Klinikum Görlitz gGmbH, Klinik für Neurochirurgie, Görlitz
  - DIAKOVERE Annastift - Orthopädische Klinik der MHH, Hanover
  - Katholisches Klinikum, Brüderhaus Koblenz, Koblenz
- Kantonsspital St. Gallen Klinik für Orthopädische Chirurgie und Traumatologie des Bewegungsapparates, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
will be decided in due time

REFERENCES:
- [Derived] Eif M, Forster T, Fleege C, Kilian F, Schmitt AD, Daentzer D. Lumbar fusion using a carbon-fiber PEEK pedicle screw system combined with a carbon-fiber PEEK TLIF cage: a prospective, multicenter study. BMC Musculoskelet Disord. 2025 Mar 6;26(1):224. doi: 10.1186/s12891-025-08457-7. PMID 40050812